CLINICAL TRIAL: NCT03844451
Title: ENHANCED RECOVERY AFTER ORTHOGNATHIC SURGERY USING LIPOSOMAL BUPIVACAINE: A RANDOMIZED CONTROL TRIAL
Brief Title: Enhanced Recovery With Liposomal Bupivacaine in Orthognathic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Kristopher Day, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-09-0046
Record Dates: First submitted 2019-01-17; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Pain, Postoperative
Keywords: Exparel, liposomal bupivacaine, postoperative, pain control
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal bupivicaine with nerve block (Experimental): The treatment group will receive an intraoperative V2 trigeminal nerve block using liposomal bupivacaine in addition to a standard bupivacaine nerve block.
  Interventions: Drug: Liposomal Bupivacaine; Drug: Bupivacaine and Epinephrine
- Nerve block only (Placebo Comparator): The control group will undergo conventional perioperative management without an ERAS protocol and standard bupivacaine intraoperative nerve block.
  Interventions: Drug: Bupivacaine and Epinephrine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — At the conclusion of the procedure, liposomal bupivacaine will be administered as a V2 nerve block.
  Arms: Liposomal bupivicaine with nerve block
Drug: Bupivacaine and Epinephrine — At the start of the procedure, 0.5% bupivacaine and 1:200,000 epinephrine as a surgical field block.

SUMMARY:
The proposed study design is a prospective, clinical trial comparing control group patients (CG; ncg = 30) that will undergo conventional perioperative management without an ERAS protocol and standard bupivacaine intraoperative nerve block to randomized treatment group patients that will receive an intraoperative V2 trigeminal nerve block using LB (TG; ntg = 30).

DETAILED DESCRIPTION:
The proposed study design is a prospective, clinical trial comparing control group patients (CG; ncg = 30) that will undergo conventional perioperative management without an ERAS protocol and standard bupivacaine intraoperative nerve block to randomized treatment group patients that will receive an intraoperative V2 trigeminal nerve block using LB (TG; ntg = 30). The total study population size (N = 60) was determined by power analysis using a free online calculator for continuous variable comparison with two-sided equality. The hypotheses for this study is that a trigeminal nerve block LB-ERAS will confer better pain control to patients undergoing OGS compared to conventional bupivacaine and no ERAS protocol. We speculate that hospital stay, pain scores, duration to first postoperative oral intake, opioid pain medication requirements, and ORAE's will all be less in the TG than the CG. We postulate that the volume of oral nutrition tolerated in the first 48-hours postoperatively will be greater in the TG than the CG. Liposomal bupivacaine will be injected after a minimum of 20 minutes have passed since the pre-operative nerve block was administered. The patients' subjective pain experienced will be quantified by a traditional 10-point visual analogue score (VAS) in the post-anesthesia care unit (PACU), at time of admission to the post-operative recovery room, throughout the inpatient recovery period, and at time of discharge. The time to tolerance of first oral intake will be measured in hours. The amount of first-48-hour oral intake will be measured in milliliters (mL). We believe that a LB-ERAS protocol will result in lower necessary doses of opioid pain medications. This will be measured as first 48-hour total mg/kg dosage of opioid pain medication converted to oxycodone-equivalents by standard conversion ratios. The incidence of ORAE's will be tallied by the number of necessary prn doses of symptomatic management anti-pyretic and anti-nausea medications. We expect this to be lower in the TG. The degree of respiratory suppression will be measured by first 48-hour respiratory rate between CG and TG patients, which we expect to be lower in the CG relative to higher opioid pain medication totals.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing orthognathic surgery at Dell Children's Medical Center will be intended for inclusion in the study.

Exclusion Criteria:

* Only those patients with insufficient data in their medical records or contraindications to the administration of liposomal bupivacaine (hepatic disease or allergy to amide local anesthetics) will be excluded from the study.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-05-17 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Duration of hospitalization status post jaw surgery | Until discharge from hospital, an average of 3 days
  The amount of time spent in the hospital after the surgery

SECONDARY OUTCOMES:
Total morphine-equivalents | First 48 hours after surgery
  Amount of morphine-equivalents consumed by patient
Pain Scores | Until discharge from hospital, an average of 3 days
  On a 1-10 visual analogue scale, measured per nursing with vital signs
Oral intake | First 48 hours after surgery
  Oral intake measured in cc

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher Day, MD, Principal Investigator — Dell Children's Medical Center of Central Texas
Locations (1):
- Dell Children's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided